CLINICAL TRIAL: NCT02971865
Title: Effect of Manual Medicine or Cognitive Behavioral Therapy With Chronic Uncontrolled Diabetes Within a Shared Primary Care Visit (A Randomized Clinical Trial)
Brief Title: Effect of Manual Medicine or Cognitive Behavioral Therapy With Chronic Uncontrolled Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Community Wellness Center, West Linn, OR (Other)
Responsible Party: Principal Investigator, Ryan Bellacov, Chairman of the board, Community Wellness Center, West Linn, OR
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000CWC
Record Dates: First submitted 2016-11-14; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Cognitive Behavior Therapy; Chiropractic; Diabetes Mellitus, Type 2; Primary care shared visit
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT/CMT (Experimental): The CBT/CMT program does not focus specifically on a particular condition such as diabetes. All treatment included patient education on nutrition content and mindfulness practice (emotions, and sensations in the present moment without trying to change them, awareness of breathing, and social economic problems) with manual therapy.
  Interventions: Behavioral: CBT/CMT
- traditional primary care visit (Active Comparator): Provide high quality primary care for men, women, and children of all ages. Our providers work together to ensure that you receive the most comprehensive care possible. Primary care is described as the medical setting in which patients receive most of their medical care and, therefore, is typically their first source for treatment
  Interventions: Other: Control group traditional primary care

INTERVENTIONS:
Behavioral: CBT/CMT — Cognitive Behavioral Therapy (CBT - training to change nutritional thoughts and behaviors) and Chiropractic Manipulative Therapy (CMT - High Velocity, low amplitude chiropractic manipulation) were delivered in average total 8 visits in a year. The interventions were comparable in format (individual visit), duration (30 minute visits), frequency (monthly), and number of participants per group (see intervention details). Each intervention was delivered according to a protocol in which all instructors were trained. (Figure 3: Chiropractic/Behavioral health and Primary care Integration Protocol.) Routine care varied with patient complaints at the time of visit.
  Other Names: Cognitive Behavioral Therapy; Chiropractic Manipulative Therapy
  Arms: CBT/CMT
Other: Control group traditional primary care — No change in care usually given
  Arms: traditional primary care visit

SUMMARY:
Effects of manual medicine or cognitive behavioral therapy with chronic uncontrolled diabetes within a shared primary care visit. An evaluation of the effectiveness of manual therapy vs cognitive behavioral therapy (CBT) vs traditional primary care visit care is in need.

DETAILED DESCRIPTION:
Integrating cognitive behavioral health nutritional therapy (hereafter CBT) and primary care services plays an important role in healthcare outcomes and the prevalence of chronic disorders treated in primary care. The Center of Disease Control has published some disturbing numbers: 9.3% of the U.S. population is affected by diabetes. Ninety-five percent of these individuals will receive treatment from their primary care provider, less than 5% will consult with a dietitian or behavioral health provider. Diabetes is projected to triple in the US despite numerous treatment options and greatly increased medical resources devoted to this problem. There is need for treatments that demonstrate an effectiveness that is low risk and wide spread.

A person's state of mind can play an important role in physical and psychosocial health conditions such as diabetes. Depression and diabetes share a bidirectional association. A recent meta-analysis reported that depressed individuals have a 60% increased risk of developing diabetes. An association was found between the risks of developing diabetes and non-severe depression, persistent depression, and untreated depression. Cognitive behavioral therapy, among others, has demonstrated effectiveness for a variety of chronic conditions.

By implementing a shared visit with primary care we encourage the advancement of this new approach. A focus on stress reduction by using mindfulness to encourage patients to think of their body as a whole and heal through not only the use of CBT, but with nutrition and manual therapy. Demonstrating the beneficial effects CBT has on uncontrolled diabetes will offer another psychosocial treatment option for the large number of suffering US residents. CBT and other mindfulness-based interventions have been recognized as helpful for a range of conditions including chronic pain. However, only 1 large randomized clinical trial (RCT) has evaluated CBT for chronic low back pain, and that trial was limited to older adults.

This clinical trial also includes chiropractic manipulative treatment (CMT) with uncontrolled diabetes patients. This study is unique due to the lack of any pre-existing trials of this nature. CMT has demonstrated improvement in physical function. A compromise of the peripheral nervous system is a common long-term complication of diabetes. In severe cases, this can lead to limb amputations and sudden cardiac death secondary to autonomic polyneuropathy. Proper recognition of the musculoskeletal manifestations of patients with diabetes will aid the treating chiropractor and alert them to the possible neurological consequences of diabetes.

ELIGIBILITY:
Inclusion Criteria:

Hemoglobin A1c above 9%

Exclusion Criteria:

* 0-18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c | One year
  lab values ([hemoglobin A1c]; range, 1-20%
Consumer Assessment of Healthcare Providers and Systems (CAHPS) | One year
  31 questions with three categories version 3.0 done at one year

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9 | One year
  PHQ-9; range, 0-27; higher scores indicate greater severity).15 The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. 14 The PHQ-9 is the depression module, which scores each of the 9 Diagnostic and Statistical Manual of Mental Disorders (DSM) -IV criteria as "0" (not at all) to "3" (nearly every day).

CONTACTS AND LOCATIONS:
Locations (1):
- Community Wellness Center, West Linn, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share individual participant data with other researchers via Journal of Manipulative and Physiological Therapeutics (JMPT). Also, annual collaborative of primary care providers in Oregon.

REFERENCES:
- [Result] Mezuk B, Eaton WW, Albrecht S, Golden SH. Depression and type 2 diabetes over the lifespan: a meta-analysis. Diabetes Care. 2008 Dec;31(12):2383-90. doi: 10.2337/dc08-0985. PMID 19033418